CLINICAL TRIAL: NCT05505929
Title: A Post-Market Registry of the BioFreedom Ultra CoCr Biolimus A9 Coated Coronary Stent System
Brief Title: eUltra 10k - Biofreedom Ultra
Status: Recruiting | Type: Observational
Sponsor: Biosensors Europe SA (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: 22-EU-01
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Post Market Clinical Follow up (PMCF)
Keywords: PMCF; Registry; Biofreedom Ultra; eUltra

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Biofreedom Ultra — The BioFreedomTM Ultra CoCr DCS is a combination product consisting of two key components: the cobalt chromium stent platform coated abluminally with the active ingredient BA9TM (polymer and carrier free) and the delivery system.

SUMMARY:
This registry captures data on BioFreedomTM Ultra CoCr DCS in standard clinical practice (real world population) and serves as Post Market Clinical Follow up (PMCF) as part of the Post-Market Surveillance.

DETAILED DESCRIPTION:
Prospective, observational multi-center registry to be conducted at up to 150 interventional cardiology centers in up to 15 countries. Patients will be followed by telephone for 1 year after PCI for data collection. This registry captures data on BioFreedomTM Ultra CoCr DCS in standard clinical practice (real world population) and serves as Post-Market Surveillance.

This registry will enroll up to 10000 patients in up to 150 investigative centers in Europe, South America, Middle East, Asia over a period of 5 years. Each patient be followed with phone (or clinic) visit at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* According to the current version of Instructions of Use (IFU)
* Patient is at least 18 years old
* Patient provides a signed informed consent

Exclusion Criteria:

* According to current version of IFU
* Patients will be excluded as per Medical Device Regulation (MDR) (Article 65: "Clinical investigations on minors" and article 66: "Clinical investigations on pregnant or breastfeeding women"
* Patients will be excluded if they are under judicial protection, guardianship or curatorship or if they are deprived of their liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational registry is open to all patients with coronary artery disease treated by percutaneous coronary intervention (PCI) with one or more BioFreedom™ Ultra CoCr DCS within the products indications of the Instructions for Use (IFU).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months

SECONDARY OUTCOMES:
Clinically driven Target Lesion Revascularization (TLR) | 12 months
Cardiovascular death (CD) | 12 months
Target Vessel MI | 12 months
Target Vessel Revascularization (TVR) | 12 months
Stent thrombosis | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Bournemouth hospital, Bournemouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided